CLINICAL TRIAL: NCT03368729
Title: A Phase 1b/2 Study of the PARP Inhibitor Niraparib in Combination With Trastuzumab in Patients With Metastatic HER2+ Breast Cancer
Brief Title: Niraparib in Combination With Trastuzumab in Metastatic HER2+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Tesaro, Inc. (Industry); Susan G. Komen Breast Cancer Foundation (Other); Breast Cancer Research Foundation of Alabama (Unknown); The V Foundation (Other)
Responsible Party: Principal Investigator, Erica Stringer-Reasor, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F2017000 (UAB 17112)
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; HER2 Positive Breast Carcinoma
Keywords: metastatic breast cancer; HER2 positive; Poly (ADP-Ribose) polymerase (PARP); Niraparib; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — niraparib; Trastuzumab

STUDY DESIGN:
Intervention Model Description: There are two phases to this study. Phase 1 will enroll 6-12 patients and Phase 2 will enroll up to 40. Trastuzumab will be given intravenously at 6 mg/kg on Day 1 for each 21 day cycle in both phases. Niraparib will be given by mouth every day at a dosage of 200 mg for phase 1 participants and 200 mg (or 100 mg) for phase 2 participants. Tumor measurement and response will be monitored by MRI or CT scans after cycles 3 and 6 and then every 12 weeks for up to 2 years or until disease progression. Blood and tissue samples will be collected for pharmacokinetics, biomarkers, and laboratory evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Niraparib 200 mg + Trastuzumab 6 mg/kg (Experimental): In phase 1 patients in this first arm will receive 200 mg Niraparib in combination with 6 mg/kg Trastuzumab given IV every 3 weeks.
  Interventions: Drug: Niraparib; Drug: Trastuzumab
- Phase 1: Niraparib 100 mg + Trastuzumab 6 mg/kg (Experimental): In phase 1 patients in this second arm will receive Niraparib 100 mg in combination with 6 mg/kg Trastuzumab given IV every 3 weeks.
  Interventions: Drug: Niraparib; Drug: Trastuzumab
- Phase 2: Niraparib 200 mg or 100 mg + Trastuzumab 6 mg/kg (Experimental): The dosage of Niraparib in phase 2 will be determined by the response of patients in Phase 1. A dosage of Niraparib 200 mg will be given along with Trastuzumab 6 mg/kg IV unless a dose limiting toxicity occurs in Phase 1. If so, Niraparib 100 mg will be given with Trastuzumab 6 mg/kg (instead of Niraparib 200 mg).
  Interventions: Drug: Niraparib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Niraparib — Niraparib is an oral PARP-1 and -2 inhibitor with high potency.
  Other Names: formerly MK-4827
Drug: Trastuzumab — Trastuzumab is a commercially available agent administered by intravenous infusion. A loading dose of 8 mg/kg will be given as the first dose followed with all subsequent doses of 6 mg/kg every 3 weeks.

SUMMARY:
The human epidermal growth factor receptor 2 (HER2) regulates cell growth and survival. Approximately 15-20% of all breast cancers are HER2-positive, which are an aggressive and fast-growing subtype of breast cancer. This study will evaluate a new treatment using a potent Poly polymerase (PARP) inhibitor known as Niraparib. Niraparib will be combined with trastuzumab, a HER2-targeted agent, to evaluate the safety and tolerability in patients with metastatic HER2 positive breast cancer. It is anticipated that the combination of drugs will improve survival and have few side effects.

DETAILED DESCRIPTION:
Treatment will be administered on an outpatient basis. All patients in the phase 1 and 2 portion of the study will receive Niraparib by mouth on days 1-21 of each 21 day cycle as well as trastuzumab intravenously (IV) on day 1 of each cycle. Blood and tissue will be collected at pre-specified times to enable pharmacokinetic, biomarker, and toxicity studies. The drug dosage will then be determined for the phase 2 portion at a dose limiting level. Following treatment, patients will be followed every 6 weeks for 6 months until disease progression or an unacceptable adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18 years
* Eastern Cooperative Oncology Group performance status 0-2 (Karnofsky >60%).
* Patients with metastatic breast cancer.
* HER2 (human epidermal growth factor receptor 2)-positive breast cancer prospectively determined on the primary tumor by a local pathology laboratory and defined as: Immunohistochemistry (IHC) score of 3+ and/or positive by ISH (defined by In Situ Hybridization ratio of ≥ 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies). Both IHC and ISH assays will be performed; however, only one positive result is required for eligibility.
* Estrogen/progesterone receptor positive OR negative disease allowed.
* Patients must have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Patients that have failed at least one anti-HER2 therapy in the metastatic setting.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mL
  * platelets ≥100,000/mL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) 5 ≤ X institutional ULN
  * creatinine ≤ institutional ULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by echocardiogram (preferred) or multigated acquisition (MUGA) scans.
* Willing and able to comply with the requirements of the protocol.
* Patient is able to take oral medication.
* Signed informed consent.
* Female patients of childbearing potential must be willing to use one highly effective form of hormonal contraception or two effective forms of nonhormonal contraception.
* Contraception must continue for the duration of study treatment and for 7 months after the last dose of study treatment. The above contraception is not a requirement in the case of any of the following:

  * The patient, or partner of the patient, is surgically sterilized.
  * The female patient is >45 years of age and is postmenopausal (has not menstruated for at least 12 consecutive months
  * The patient truly abstains from sexual activity and when this is the preferred option to avoid conception and contraception and/or usual lifestyle of the patient.

Exclusion Criteria:

* Metastatic breast cancer patients who are HER2 positive and have NOT progressed on at least one prior HER2-targeted therapies for metastatic disease
* Patients who have not recovered from CTCAE, v. 4.03 grade 2 or higher toxicities of prior therapy to the point that they would be appropriate for re-dosing will be ineligible for study treatment. Subjects receiving weekly therapy must have a washout period from prior chemotherapy of as least one week. Washout period for chemotherapy administered every 2, 3, or 4 weeks will be 2, 3, and 4 weeks respectively, provided subject has recovered from toxicities of prior therapy such that retreatment is appropriate.
* Patients must be at least two weeks from prior RT
* Patients must have a one-week washout period from prior hormonal therapy (e.g. testosterone, estrogen, progestin, gonadotropin-releasing hormone antagonist).
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not been using steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.

No concurrent anti-cancer treatment of any type

* Patients with known germline BRCA 1 or BRCA 2 mutations
* Patient has undergone prior treatment with a known poly(ADP-ribose) polymerase (PARP) inhibitor.
* Prior treatment of a total doxorubicin >360 mg/m2 (or equivalent)
* Patient has known active hepatitis B (eg, hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (eg, hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected).
* Patient has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Chronic immunosuppressive therapies including systemic corticosteroids or concurrent short-term use of immunosuppressive therapies is not allowed. Short- term corticosteroid use must be discontinued at least 2 weeks prior to study treatment.
* Patients with known grade 2 or greater allergic reactions attributed to compounds of similar chemical or biological composition to niraparib are ineligible for study enrollment.
* Patients with known grade 2 or greater allergic reactions attributed to compounds of similar chemical or biological composition to herceptin are ineligible for study enrollment.
* Patient is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of study treatment.
* History of non-breast malignancies within the 5 years prior to study entry, except for the following:

  * Carcinoma in situ (CIS) of the cervix
  * CIS of the colon
  * Melanoma in situ
  * Basal cell and squamous cell carcinomas of the skin
* Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active infection that requires systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
* Cardiopulmonary dysfunction as defined by any of the following prior to randomization:

  * History of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.0) Grade ≥3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) criteria Class ≥ II
  * Angina pectoris requiring anti-angina medication, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease
  * High-risk uncontrolled arrhythmias (i.e. atrial tachycardia with a heart rate >100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block [second degree AV-block Type 2 [Mobitz 2] or third degree AV-block])
  * Significant symptoms (Grade ≥2) relating to left ventricular dysfunction, cardiac arrhythmia, or cardiac ischemia
  * Myocardial infarction within 12 months prior to randomization
  * Uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg)
  * Evidence of transmural infarction on ECG
  * Heart-rate corrected QT interval (QTc) prolongation >470 msec at screening.
  * Requirement for oxygen therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for women only.
Enrollment: 46 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-limiting toxicity (DLT) | Baseline to 6 weeks
  A DLT is defined as hematological events > or equal to grade 3 leukopenia, anemia, and thrombocytopenia and also non-hematological events > or equal to grade 3 fatigue, nausea, constipation, vomiting, or diarrhea.
Phase 2: Objective Response Rate | Baseline up to 100 weeks
  Response and progression of disease will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Committee.

SECONDARY OUTCOMES:
Number of adverse events | Baseline up to 100 weeks
  Toxicities will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) v. 4.03.
Progression-free survival | Baseline to the date of first documented progression to date of death from any cause, whichever comes first, assessed up to 100 months
  The RECIST v. 1.1 criteria will be used to evaluate progression-free survival as well as CT and MRI scans. Progression is indicative of existing target and non-target lesions.
Phase 1: Niraparib levels | Baseline to 25 days
  Plasma niraparib levels will be assessed at specific time points in participants blood during cycle 2 treatment in Phase I patients only. A population pharmacokinetic modeling approach will be used to describe area under the curve (AUC) plasma concentrations of niraparib and its metabolites in participants in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Stringer-Reasor, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington-, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No